CLINICAL TRIAL: NCT07069361
Title: The Role of Mindful Emotion Regulation in Organizational Contexts: A Workplace Experiment
Brief Title: Mindful Emotion Regulation in Organizational Contexts
Acronym: MEROC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bucharest (Other)
Responsible Party: Principal Investigator, Cezar Giosan, Associate Professor of Psychology, University of Bucharest
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 008
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Mindfulness Based Cognitive Therapy; Wait-List Control; Emotion Regulation; Organizational Context
Keywords: Mindfulness; Mindfulness for Life; Intervention; Emotion Regulation; Organizational Outcomes; Randomized Controlled Trial
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This study uses a two-period crossover design. Participants are randomly assigned to one of two sequences: (1) immediate intervention with Mindfulness-Based Cognitive Therapy for Life (MBCT-L) followed by a no-treatment follow-up period, or (2) initial wait-list control with no intervention followed by MBCT-L. Each phase lasts 8 weeks, with outcome assessments conducted at the end of each phase. The baseline measurement preintervention is in the week preceding the start of the first phase of the study.This design allows for both between-group comparisons during the first phase and within-subject comparisons across the two phases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness-Based Cognitive Therapy - Life Course Adaptation (MBCT-L) (Experimental): Mindfulness For Life (MBCT-L) is an adapted version of Mindfulness-Based Cognitive Therapy, designed for the general population. While rooted in the original MBCT program, which was developed for preventing depressive relapse, Mindfulness for Life is tailored to increase the levels of psychological well-being, emotional resilience and mental health outcomes in non-clinical populations.
  The program consist of 8 weekly sessions of 2 hours and 15 minutes, complemented by guide daily home practice. Participants are taught mindfulness meditation practices, cognitive-behavioral strategies, and experiential exercises aimed at enhancing self-awareness and emotional regulation. The intervention follows the standardized 'Mindfulness for Life' curriculum, as developed by the Oxford Mindfulness Foundation (OMF), and is delivered by an instructor trained in the approach through OMF.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy - Life Course Adaptation (MBCT-L)
- Wait-List Control Group (No Intervention): Participants in the wait-list control group will not receive the intervention during the initial study period but will be offered access to the Mindfulness for Life (MBCT-L) program after the initial phase of the study ends. For the first 8 weeks, they will not receive any structured psychological intervention as part of the study. They will continue any usual care or personal routines, an they will complete the same assements at equivalent time points.
  After this initial waiting period and completion of the first follow-up assessment, participants will then begin the Mindfulness for Life (MBCT-L) program.
- Wait-List Control Group Phase 2 (No Intervention): This is the second phase of a two-period crossover study. During this phase, participants assigned to the wait-list control condition do not receive any psychological intervention or active treatment. They continue with their usual activities and complete outcome assessments. In Phase 1 of the trial, the participants assigned to this group received the MBCT-L interventions.
- Mindfulness for Life - Mindfulness- Based Cognitive Therapy Adaptation (MBCT-L) Phase 2 (Experimental): This is the second phase of a two-period crossover study. During this phase, participants who were originally assigned to the wait-list control group now receive the MBCT-L intervention.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy - Life Course Adaptation (MBCT-L)

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy - Life Course Adaptation (MBCT-L) — MBCT-L (Mindfulness-Based Cognitive Therapy for Life) Is a structered, group-based intervention developed for use with healthy adults. The programs runs for 8 consecutive weeks, with sessions lasting 2 hours and 15 minutes. It includes formal and informal mindfulness practices, exercises to develop cognitive and emotion awareness, with elements adapted from cognitive therapy. The course was designed to support participants in cultivating habits that increase emotion regulation and psychological well-being. Home practice is assigned daily using audio-guided meditations. The intervention is standardized and delivered by a instructor trained under Oxford Mindfulness Centre (OMC) protocols. MBCT-L is distinct from the clinical MBCT model used for relapse prevention. And it is also disting from other Mindfulness-Based interventions as it uses different exercises than, for example, Mindfulness-Based Stress Reduction which emphasis stress theories in the intervention.
  Arms: Mindfulness for Life - Mindfulness- Based Cognitive Therapy Adaptation (MBCT-L) Phase 2; Mindfulness-Based Cognitive Therapy - Life Course Adaptation (MBCT-L)

SUMMARY:
This randomized controlled trial investigates the effects of an 8-week mindfulness-based interventions, Mindfulness for Life (MBCT-L) on daily emotion regulation, psychological functioning, and work-related outcomes. The primary objective of this study is to investigate the underlying mechanism of change between mindfulness and job performance and satisfaction.

DETAILED DESCRIPTION:
This study investigates the mechanisms by which mindfulness training influences positive affect, job performance, and satisfaction in organizational settings. Employing a two-period crossover design, participants receive an 8-week Mindfulness for Life (MBCT-L) intervention. Guided by Mindfulness-to-Meaning theory, the investigator propose that increases in mindfulness enhance positive affect through improved decentering and positive reframing. In line with the Broaden-and-Build theory, it is hypothesized that heightened positive affect leads to better in-role job performance and higher job satisfaction by increasing psychological capital. The primary objective is to elucidate these mediational pathways, thereby advancing our understanding of how mindfulness interventions can foster improve emotion regulation and organizational functioning.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Full-time Workers

Exclusion Criteria:

* Experiencing Hallucinations
* Experiencing psychotic symptoms
* Recieving psychotropic medications
* Experiencing legal or health issues that would prevent them to attend the sessions.
* Have had participated in a Mindfulness-Based course in the last 2 years.
* Presenting symptoms of intellectual disability, communication disorders or neurocognitive disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2025-07-30 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Multidimensional State Mindfulness Questionnaire (MSMQ) | Baseline (pre-intervention), week 8 (post-first phase), and week 16 (end of study following crossover).
  This scale is used to measure daily changes in state mindfulness. Participants will self-report levels of acting with awareness, nonjudgemental acceptance and present-moment attention in the context of their work day. The Multidimensional State Mindfulness Questionnaire (MSMQ) includes 9 items, rated on a Likert-type scale, and is designed to capture mindfulness as it fluctuates over time. Data will be collected across three daily diary periods: a baseline period before any intervention, a second period following the first 8-week phase, and a final period conducted after the second 8-week phase, once the crossover is complete. This structure allows for the examination of both between-group and within-subject changes in state mindfulness associated with the intervention.

SECONDARY OUTCOMES:
Metacognitive Processes of Decentering - State Scale (MPoD-s) | Baseline (pre-intervention), week 8 (post-first phase), and week 16 (end of study following crossover)
  The Metacognitive Processes of Decentering is a brief self-report measure designet to assess momentary decentering. The capacity to observe thoughts and emotions with perspective and distance from one's experience. The current implementations includes two items: "I can watch my thoughts and emotions come and go like clouds" and "I am more than my thoughts and feelings," rated on a Likert scale. The third decentering item was omitted to preserve conceptual compatibility with related constructs. The scale will be used in three periods of daily diary thought the study, first one after interventions, post-interventions phase 1, and at the end of the study after the crossover is complete.
Positive Reframing | Baseline (pre-intervention), week 8 (post-first phase), and week 16 (end of study following crossover)
  We used the Positive Reframing subscale from the Brief COPE inventory to assess participants' tendency to reinterpret challenging situations in a more constructive or optimistic way. This subscale includes two items rated on Likert scale. This scale is part of the daily dairies.
Positive and Negative Affect Schedule - Short Form (PANAS-SF) | Baseline (pre-intervention), week 8 (post-first phase), and week 16 (end of study following crossover).
  PANAS-SF is a 20 item self-report measure used to assess two distinct dimensions of affect: positive affect and negative affect. The instructions to this questionnaire were adapted to a daily level. Participants were instructed to think about the affects they experienced through their work day. They rate the extent to which they have experienced specific emotions in the workplace today. This scale is part of the daily diaries.
Psychological Capital | Baseline (pre-intervention), week 8 (post-first phase), and week 16 (end of study following crossover)
  Psychological Capital Questionnaire (PCQ-12) is the short version of PCQ-24. It measures four core components of psychological capital: hope (4 items), self-efficacy (3 items), resilience (3 items), and optimism (2 items). Each item is rated on a 6-point Likert scale. This scale is included in the daily diaries.
In-Role Job Performance | Baseline (pre-intervention), week 8 (post-first phase), and week 16 (end of study following crossover)
  In-role job performance was assessed using a 7-item scale developed by Williams and Anderson (1991), designed to measure how well employees fulfill the formal requirements of their job as outlined in their job description. Respondents rate items reflecting task completion, responsibility fulfillment, and expected work duties (e.g., "I perform tasks that are expected of me," "I meet the formal requirements of my job") using a Likert-type scale. This was adapted to a daily level and included in the diaries.
Short Index of Job Satisfaction (SIJS) | Baseline (pre-intervention), week 8 (post-first phase), and week 16 (end of study following crossover)
  The Short Index of Job Satisfaction (SIJS) is a brief, 5-item self-report instrument designed to assess global job satisfaction. Respondents rate each item on a 5-point Likert scale ranging from 1 ("strongly disagree") to 5 ("strongly agree"), with higher scores indicating greater overall satisfaction with one's job. The SIJS captures a unidimensional construct of job satisfaction and it has been adapted to a daily level. This scale was included in the daily diaries.
Single Item Sleep Quality Scale | Baseline (pre-intervention), week 8 (post-first phase), and week 16 (end of study following crossover)
  This scale is a brief self-report measure designed to assess overall sleep quality. It uses a Likert scale from 0 to 10, where 0 represents the worst posible sleep and 10 the best of quality. This scale has favorable measurement characteristics similar to Pittsburgh Sleep Quality Index (PSQI). It is used in the daily diaries of this study.
Substance Use | Baseline (pre-intervention), week 8 (post-first phase), and week 16 (end of study following crossover)
  Substance Use subscale is used from the Brief COPE inventory o assess the extent to which participants use alcohol or other substances as a coping strategy in response to stress. This subscale consists of two items rated on a Likert scale. In addition, we included three single-item questions to capture actual substance consumption: "How many cigarettes did you smoke yesterday?", "How many doses of alcohol did you consume yesterday?" (e.g., one 330 ml beer, one 150 ml glass of wine, or one 40 ml shot of spirits), and "Did you use any other substances that could alter your state of consciousness?" These items were designed to provide a more detailed, behaviorally anchored assessment of substance use on a daily basis. This scale is included in the daily diaries.
Single-item Emotion Regulation Strategies | Baseline (pre-intervention), week 8 (post-first phase), and week 16 (end of study following crossover)
  A set of five single-item measures is included to assess key emotion regulation strategies in a daily context. Each item targeted a specific strategy: active coping ("I took active steps to improve the situation"), attention distraction ("I distracted myself from the situation or my feelings"), rumination ("I thought repeatedly about the situation or my feelings"), cognitive reappraisal ("I tried to change my perspective on the situation or change how I think about it"), and emotional suppression ("I held back from expressing my emotions"). Respondents rated each item on a Likert-type scale reflecting the extent to which they used that strategy on a given day. This items were included in the daily diaries.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bucharest, Bucharest, Sector 5, Romania

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 1 January 2026 to 1 January 2031

REFERENCES:
- [Background] Hanley AW, de Vibe M, Solhaug I, Farb N, Goldin PR, Gross JJ, Garland EL. Modeling the mindfulness-to-meaning theory's mindful reappraisal hypothesis: Replication with longitudinal data from a randomized controlled study. Stress Health. 2021 Oct;37(4):778-789. doi: 10.1002/smi.3035. Epub 2021 Mar 9. PMID 33607697
- [Background] Wang Y, Garland EL, Farb NAS. An experimental test of the mindfulness-to-meaning theory: Casual pathways between decentering, reappraisal, and well-being. Emotion. 2023 Dec;23(8):2243-2258. doi: 10.1037/emo0001252. Epub 2023 May 11. PMID 37166828